CLINICAL TRIAL: NCT03859622
Title: CYP2D6 Polymorphism Defining UM, IM, NM and PM Status in Unselected Medically Treated Patients of General Practice in Austria
Brief Title: CYP2D6 Polymorphism in Patients of General Practice in Austria
Status: Completed | Type: Observational
Sponsor: Karl Landsteiner Institute for Systematics in General Medicine (Other)
Responsible Party: Principal Investigator, Gustav Kamenski, General Practitioner/Family Physician, Karl Landsteiner Institute for Systematics in General Medicine
Other Study IDs: KarlLandsteinerISGM CYP2D6
Record Dates: First submitted 2018-10-20; First posted 2019-03-01 (Actual); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Disorder Due Cytochrome P450 CYP2D6 Variant
Keywords: Cytochrome P 450 CYP2D6 Variants; Genetic polymorphism; Practice, Family; Drug metabolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA extraction from peripheral white blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CYP 2D6 enzyme metabolizes a significant number of drugs frequently prescribed in general practice/ family medicine. Various genetically different variants define if the patient is an ultra-rapid (UM), an normal (NM) (the normal case), an intermediate (IM) or a poor metabolizer (PM). It is estimated that approximately 20- 25 % of frequently described drugs are activated to more active or metabolized to ineffective or less effective drugs by CYP 2D6. Substrates of CYP 2D6 are mainly antidepressants, neuroleptics, opioids (e.g. codeine), beta-blockers, anti-arrhythmic drugs and various other single drugs. In case of an UM a drug can be metabolized too rapidly losing its therapeutic effect, requiring a higher dosage, or it can have a toxic effect, if it is converted too rapidly in the effective form (e.g. codeine). If metabolized too slowly (PM) it can accumulate and reach toxic levels.

In this observational study (1) data relating to the number of patients of a single Austrian general practice receiving one or more drugs metabolized by CYP 2D6 are collected by extracting their electronic records of the last 3 years. In addition (2) consecutive patients with unknown genetic status of their CYP 2D6 enzyme visiting the surgery for a routine blood test due to various reasons, are additionally tested for their CYP 2D6 metabolizing status, if they actually take a drug metabolized by CYP 2D6.

The aim of the study is to generate CYP 2D6 polymorphism data from Caucasian patients of an average Austrian general practice for the first time, which allows to group patients according to their NM, UM, IM and PM status. This can be of considerable clinical relevance when prescribing specific drugs. This study tries to investigate in how many patients the knowledge of the CYP 2D6 metabolizing status could have an influence on choosing the actually prescribed drug. In addition we plan to describe the distribution of frequent and relevant CYP 2D6 alleles including their combinations in patients of an average Austrian general practice for comparison reasons with other Caucasian populations.

DETAILED DESCRIPTION:
Study population:

Unselected consecutive patients of the practice office visiting the surgery for a routine blood sampling due to various medical conditions and who are prescribed or have been prescribed drugs metabolized by the CYP2D6 enzyme (or drugs being a strong inhibitor of CYP 2D6) during the last 3 years. Only in these patients CYP2D6 polymorphism is determined using a fraction of the EDTA-blood sample. No further genetic investigations or additional blood collections are performed.

Patients who are considered to be eligible to participate in the study have to sign an informed consent after being informed about the aims of the study.

Blood sampling and processing of the specimens:

A standardized blood sampling using a Vacutainer system with filling of an EDTA tube (4 ml) for the red and white blood count is performed. 300 microliters of the collected blood are used for further determination of the CYP2D6 polymorphism.

Isolation of DNA:

DNA is extracted from EDTA blood in the practice laboratory by using the Spin Micro Extraction Kit® (ViennaLab,Vienna). The concentration and quality of DNA is measured using a Bio Photometer plus (Eppendorf). The extracted DNA is stored at -81°C in an ultra-low temperature deep freezer (U101-86, New Brunswick Scientific Co., Inc) without any further additives.

Real-time PCR for determination of copy number of the CYP2D6 gene:

For the determination of the copy number of the CYP2D6 gene a real-time PCR in triplicates on an ABI StepOnePlus by using the CYP2D6 RealFast™ CNV Assay (ViennaLab) is performed in the practice laboratory.

The test is based on the fluorogenic 5' nuclease assay, also known as TaqMan® assay. Each reaction contains gene-specific primer pairs for amplification of CYP2D6 and endogenous control (EC) gene fragments with 141 bp each. Further components are two dual-labeled, gene-specific hydrolysis probes, the FAM-labeled CYP2D6 probe and the HEX-labeled EC probe, which hybridize to an internal sequence of the amplified fragments. The proximity of the 5'-fluorescent reporter and 3'-quencher dye on intact probes prevents the reporter from fluorescing. During the extension phase of PCR the 5' - 3' exonuclease activity of Taq DNA polymerase cleaves the 5'-fluorescent reporter from the hybridized probe. The physical separation of the fluorophore from the quencher dye generates a fluorescent signal in real-time, which is proportional to the accumulated PCR product. The CYP2D6 RealFast™ CNV Assay is a relative quantitation assay and compares the amount of both nucleic acid targets (CYP2D6 and EC) in relation to the CYP2D6 CNV Calibrator. The EC gene is used to normalize fluorescence signals between different samples and serves as a PCR positive control.

For additional normalization of data ROX dye to a final concentration of 1 microliter to the 2 x Probe Mix is added.

RT- PCR cycling conditions for the ABI StepOneplus cycler: Initial denaturation: 95°C 10 min 1 cycle; denaturation 95°C 15 sec 40 cycles; annealing /extension 60°C 1 min.

PCR and hybridisation for CYP2D6 allele determination by the PGX-CYP2D StripAssay™:

This assay is used for a subset of samples in this study and covers only 3 polymorphic loci: 1795delT (2D6*6), 1934G>A (2D6*4) and 2637delA (2D6*3). The test principle and procedure are similar to the PGX-CYP2D6 XL StripAssay® as described below but using different cycling conditions for the Palm-Cycler (Corbett Life Science): pre-PCR: 94°C/2 min; thermocycling: 94°C/15 sec.- 58°C/ 30 sec.-72°C/30 sec (35 cycles); final extension: 72°C/3 min.

PCR and hybridisation for CYP2D6 allele determination by the PGX-CYP2D6 XL StripAssay®:

For the determination of 19 clinically relevant CYP2D6 alleles (*1; *2 A, *2 B-M; *3, *4A-H, K, L or P, *4J or N, *4M; *5; *6 A, B or D, *6C; *7, *8; *9,; *10A or B, *10 C or D; *11; *12; *14; *15; *17; *29; *35; *39; *40 or *58; *41) a PCR amplification on a Palm-Cycler (Corbett Life Science, Eight Mile Plains, QLD 4113, Australia) using biotinylated primers is first performed. The amplification products are further hybridized to a test strip containing allele-specific oligonucleotide probes immobilized as an array of parallel lines. Bound biotinylated sequences are detected using streptavidin-alkaline phosphatase and color substrates. The evaluation of this reaction is done manually by using the StripAssay®-Evaluator (ViennaLab,Vienna), a proprietary PC program to determine the homozygous or heterozygous genotype.

Cycling conditions for the Palm-Cycler (Corbett Life Science): pre-PCR: 95°C/4 min; thermocycling: 95°C/25 sec.- 60°C/ 45sec.-72°C/1min (36 cycles); final extension: 72°C/3 min.

Statistics:

The data were recorded and analyzed using Microsoft Excel Version 10 and the R Language and Environment for Statistical Computing and Graphics, Version 2.9. Standard methods are used for the description of data (frequencies and percentages for categorical data, mean and standard deviation for continuous data). To compare frequencies of CYP2D6-specific drugs prescribed in the single practice with the total number of the respective prescriptions in Lower Austria, Spearman's rank correlation-coefficient is calculated. Differences between groups were calculated by paired t-test. A p-value < 0.05 was considered to indicate statistical significance.

The Hardy-Weinberg- equilibrium was calculated using Fisher´s Exact Chi-Square test due to the small numbers of genotypes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of hypertension, diabetes, chronic heart failure, hyperlipidemias, depression, schizophrenia, cardial arrhythmias, thyroid diseases and dementia

Exclusion Criteria:

* acute infectious diseases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected consecutive patients of an Austrian general practice suffering from chronic diseases visting the practice office for a routine blood test
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Kamenski, Principal Investigator — Karl Landsteiner Institute for Systematics in General Medicine
Locations (1):
- Practice Office, Angern, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: Yes
Distribution of CYP 2D6 polymorphism and CYP 2D6 metabolizer- status (based on allele combination and copy number Variation) can be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2018 and 2019
Access Criteria: Researchers working in the pharmacogenetic field

REFERENCES:
- [Derived] Kamenski G, Ayazseven S, Berndt A, Fink W, Kamenski L, Zehetmayer S, Puhringer H. Clinical Relevance of CYP2D6 Polymorphisms in Patients of an Austrian Medical Practice: A Family Practice-Based Observational Study. Drugs Real World Outcomes. 2020 Mar;7(1):63-73. doi: 10.1007/s40801-019-00177-4. PMID 31863305

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational Cohort Cross-sectional Study: The study takes place in an average Austrian general practice in 2017 and 2018 enrolling 289 unselected consecutive patients visiting the practice office for a routine blood test for various chronic medical conditions. Only in case a patient is actually taking or has been prescribed a drug metabolized by CYP2D6 (or a drug which is a strong inhibitor of CYP2D6) within the last 3 years, the genetic polymorphism of CYP2D6 is determined. No further genetic investigations, additional blood collections or interventions are performed.
Period: Overall Study
Arm/Group | Observational Cohort Cross-sectional Study
Started | 289
Completed | 289
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Observational Cohort Cross-sectional Study: The study takes place in an average Austrian general practice in 2017 and 2018 enrolling 289 unselected consecutive patients visiting the practice office for a routine blood test for various chronic medical conditions. Only in case a patient is actually taking or has been prescribed a drug metabolized by CYP2D6 (or a drug which is a strong inhibitor of CYP2D6) within the last 3 years, the genetic polymorphism of CYP2D6 is determined. No further genetic investigations, additional blood collections or interventions are performed. All participants gave written consent.
Arm/Group | Observational Cohort Cross-sectional Study
Number analyzed (Participants) | 289
Age, Categorical [Count of Participants; unit: Participants] — Population: Baseline: 289 participants
  Participants
    <=18 years | 0
    Between 18 and 65 years | 90
    >=65 years | 199
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 289
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — In this observational study, performed in an average Austrian General Practice, the baseline distribution of alleles, genotypes and metabolizer types was determined.
  This analysis is performed for each of the 289 participants.
  Participants
    Austria | 289
Number of patients with a prescription of a CYP2D6 specific drug and routine blood test [Count of Participants; unit: Participants] — 289 consecutive participants who had a prescription of a CYP2D6 specific drug at least once within the past 3 years and who are visiting the practice during the study period of one year (2017-2018) for a planned routine blood test are tested for their different CYP2D6 alleles, genotypes and metabolizer status (PM,IM, NM, UM) in addition.
  Participants | 289

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Metabolizer Status (PM, IM, NM, UM) in Patients
Description: Remark: each participant possesses a) two individual CYP2D6 alleles, b) from the combination of these two alleles one individual genotype is derived and c) from this genotype the genetically determined metabolizer status (PM, IM, NM, UM) is derived.
  A patient can be considered a ultra-rapid (UM), a normal (NM), an intermediate (IM), or a poor metabolizer (PM) of a given drug
Time Frame: 1 Year
Population: 289 unselected consecutive patients with a prescription of a CYP2D6 relevant drug during the last 3 years and who are visiting the practice office for a routine blood test. Due to technical problems the metabolizer status of two patients could not be determined!
Measure: Count of Participants; unit: Participants
Groups:
- Frequencies of Metabolizer Status (PM, IM, NM, UM): In 289 unselected consecutive patients visiting the practice office for a routine blood test for various chronic medical conditions and only in case the patient has been prescribed a drug metabolized by the CYP2D6 enzyme (or a drug which is a strong inhibitor of CYP2D6) within the last 3 years, his or her metabolizer status (PM,IM,NM, UM) is analysed.
Arm/Group | Frequencies of Metabolizer Status (PM, IM, NM, UM)
Number analyzed (Participants) | 287
Participants
  Normal Metabolizer (NM) | 233
  Poor Metabolizer (PM) | 22
  Intermediate Metabolizer (IM) | 21
  Ultra-rapid Metabolizer (UM) | 11
Statistical Analysis 1: Comparison: Frequencies of Metabolizer Status (PM, IM, NM, UM); Standard methods are used for the description of data (frequencies and percentages for categorical data); Test type: Other — Frequencies and percentages for categorical data; Standard methods are used for the description of data (frequencies and percentages for categorical data); Standard methods are used for the description of data (frequencies and percentages for categorical data)

2. Primary Outcome: Frequency of CYP2D6 Alleles in Patients
Description: The frequency of 19 different CYP2D6 alleles in 287 patients is determined. In 2 out of all 289 patients the determination was not possible due to technical problems.
  Remark: each participant possesses a) two individual CYP2D6 alleles, b) from the combination of these two alleles one individual genotype is derived and c) from this genotype the genetically determined metabolizer status (PM, IM, NM, UM) is derived.
Time Frame: 1 Year
Population: In 289 unselected consecutive patients visiting the practice office for a routine blood test for various chronic medical conditions and only in case the patient has been prescribed a drug metabolized by the CYP2D6 enzyme (or a drug which is a strong inhibitor of CYP2D6) within the last 3 years, his or her CYP2D6 alleles are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Cohort Cross-sectional Study
Number analyzed (Participants) | 287
Participants
  *1s | 55
  *4s | 25
  *6s | 7
  *5s | 5
  *3s | 3
  *1 | 122
  *4A-H,K,L or P | 80
  *2A | 77
  *41 | 26
  *35 | 30
  *5 | 18
  *9 | 12
  *10A or B | 9
  *3 | 8
  *6A,B or D | 7
  *39 | 1
  *2B-M | 1
  *17 | 1
  *15 | 1

3. Primary Outcome: Frequency of CYP2D6 Genotypes in Patients
Description: The frequency of 61 different CYP2D6 genotypes in 287 patients is determined. In 2 out of all 289 patients the determination was not possible due to technical problems.
  Remark: each participant possesses a) two individual CYP2D6 alleles, b) from the combination of these two alleles one individual genotype is derived and c) from this genotype the genetically determined metabolizer status (PM, IM, NM, UM) is derived.
Time Frame: 1 Year
Population: 289 unselected consecutive patients with a prescription of a CYP2D6 relevant drug during the last 3 years and who are visiting the practice office for a routine blood test. Due to technical problems the genotypes of two patients could not be determined!
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Cohort Cross-sectional Study
Number analyzed (Participants) | 287
Participants
  *1s/*1s | 23
  *1s/*4s | 19
  *1s/*6s | 5
  *1s/*5s | 3
  *1s/*1s xN | 2
  *4s/*5s | 2
  *1s/*4s xN | 2
  *1s/*3s | 1
  *4s/*6s | 1
  *3s/*6s | 1
  *3s/*4s | 1
  *1/*2A | 29
  *1/*4A-H,K,L or P | 25
  *1/*1 | 24
  *2A/*4A-H,K,L or P | 15
  *1/*41 | 11
  *4A-H,K,L or P/*4A-H,K,L or P | 10
  *4A-H,K,L or P/*41 | 9
  *1/*5 | 9
  *2A/*2A | 7
  *4A-H,K,L or P/*35 | 6
  *1/*35 | 6
  *2A/*35 | 5
  *4A-H,K,L or P/*9 | 4
  *35/*41 | 4
  *2A/*41 | 4
  *1/*10A or B | 4
  *4A-H,K,L or P/10A or B | 3
  *4A-H,K,L or P/*6A,B or D | 3
  *41/*41 | 3
  *2A/*5 | 3
  *1/*3 | 3
  *9/*41 | 2
  *9/*35 | 2
  *5/*41 | 2
  *4A-H,K,L or P/*5 | 2
  *2A/*9 | 2
  *2A/*35 xN | 2
  *2A/*2A xN | 2
  *1/*9 | 2
  *1/*6A,B or D | 2
  *1/*2A xN | 2
  *1/*1 xN | 2
  *6A, B or D/*41 xN | 1
  *5/*5 | 1
  *5/*35 | 1
  *35/*39 | 1
  *35/*35 | 1
  *3/*4A-H,K,L or P | 1
  *3/*41 | 1
  *3/*10A or B | 1
  *2A/*4A-H,K,L or P xN | 1
  *2A/*3 xN | 1
  *2A/*3 | 1
  *2A/*2B-M | 1
  *2A/*10A or B | 1
  *2A/*17 | 1
  *15/*35 xN | 1
  *1/*6A,B or D xN | 1
  *1/*4A-H,K,L or P xN | 1
  *1/*35 xN | 1

4. Secondary Outcome: Number of Participants in Whom the Family Physician Considered Prior Knowledge of Their Metabolizer Status Important Before the CYP2D6-specific Drug Was Prescriped.
Description: In how many patients would family physician's knowledge of the CYP 2D6 metabolizer status (ultrarapid (UM), normal (NM), intermediate (IM) and poor (PM)) have been of importance before prescribing a CYP2D6 specific drug. Remark: The relevant drug has already already been prescribed before analysis has been taken place.
Time Frame: 1 Year
Population: 289 unselected consecutive patients with a prescription of a CYP2D6 relevant drug during the last 3 years visiting the practice office for a routine blood test. Due to technical problems only 287 could be analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Relevant Knowledge of Metabolizer Status: In 287 unselected consecutive patients visiting the practice office for a routine blood test for various chronic medical conditions and only in case the patient has been prescribed a drug metabolized by the CYP2D6 enzyme (or a drug which is a strong inhibitor of CYP2D6) within the last 3 years, it was analyzed, if physician's knowledge of his or her metabolizer status would have been of relevance before prescribing the drug.
Arm/Group | Patients With Relevant Knowledge of Metabolizer Status
Number analyzed (Participants) | 287
Participants | 29

5. Secondary Outcome: Specific Number of Patients of the Whole Practice Population Whose Electronic Health Records (EHRs) Were Assessed.
Description: The specific number of participants of the practice population with a prescription of drugs metabolized by CYP 2D6 within the last 3 years. These data were extracted from the electronic health records (EHRs) of the practice office. For this data extraction enrollement in the study and signing an informed consent was not necessary. No other data (i.e. baseline assessments, other outcome measures and adverse events) were collected in this group.
Time Frame: 1 Year
Population: Specific number of participants of the whole practice population with a prescription of a CYP2D6 relevant drug. Participants belonging to this specific group did not need to sign an informed consent form. No other data (i.e. baseline assessments, other outcome measures and adverse events) were collected in this group.
Measure: Count of Participants; unit: Participants
Groups:
- Specific Number of Patients Prescribed a CYP2D6 Relevant Drug: This secondary outcome measure serves to find out how many patients of the whole practice population got at least one prescription of an CYP2D6 metabolized drug (or an inhibitor of CYP2D6) within the last 3 years. The data were extracted from the electronic health records of the practice office. These data have only importance for pharmaco-epidemiological considerations.
Arm/Group | Specific Number of Patients Prescribed a CYP2D6 Relevant Drug
Number analyzed (Participants) | 3016
Participants | 668

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Observational Cohort Cross-sectional Study: The study takes place in an average Austrian general practice in 2017 and 2018 enrolling 297 unselected consecutive patients visiting the practice office for a routine blood test for various chronic medical conditions. Only in case a patient is actually taking or has been prescribed a drug metabolized by CYP2D6 (or a drug which is a strong inhibitor of CYP2D6) within the last 3 years, the genetic polymorphism of CYP2D6 is determined. No further genetic investigations, additional blood collections or interventions are performed.
Arm/Group | Observational Cohort Cross-sectional Study
All-Cause Mortality (participants affected / at risk) | 0/289
Serious Adverse Events (participants affected / at risk) | 0/289
Other Adverse Events (participants affected / at risk) | 0/289

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT03859622/Prot_SAP_000.pdf